CLINICAL TRIAL: NCT04862234
Title: Perioperative Stress Hyperglycemia in General and Vascular Surgery Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This clinical trial was terminated on June 7, 2024 due to new information about contraindications of using the study drug in this population.
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Georgia Davis, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00097659; K23DK122199 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Hyperglycemia Stress
Keywords: Perioperative; Surgery; Stress Hyperglycemia
MeSH Terms: interventions — dulaglutide; Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dulaglutide (Experimental): Participants randomized to receive dulaglutide within 72 hours prior to a planned surgery.
  Interventions: Drug: Dulaglutide; Device: Continuous glucose monitor (CGM), blinded
- Placebo (Placebo Comparator): Participants randomized to receive a placebo to match dulaglutide within 72 hours prior to a planned surgery.
  Interventions: Drug: Placebo; Device: Continuous glucose monitor (CGM), blinded

INTERVENTIONS:
Drug: Dulaglutide — A subcutaneous injection of dulaglutide 0.75 mg will be administered within 72 hours prior to a planned surgical intervention.
  Other Names: Trulicity
  Arms: Dulaglutide
Drug: Placebo — A subcutaneous injection of a saline placebo will be administered within 72 hours prior to a planned surgical intervention.
  Arms: Placebo
Device: Continuous glucose monitor (CGM), blinded — Continuous glucose monitor (CGM) sensor will be placed preoperatively and continued during surgical hospitalization to monitor glucose levels. CGM provides an estimated capillary blood glucose (BG) level through direct measurement of interstitial glucose levels every 5-15 minutes.
  Other Names: FreeStyle Libre Pro

SUMMARY:
Hyperglycemia is seen in approximately 30% of patients who do not have a history of diabetes and undergo general surgery. Hyperglycemia in this setting is associated with increased risk of postoperative complications. The purpose of this study is to investigate risk factors for developing high sugars during the time of surgery, and if these high sugars can be prevented by the use of an injectable diabetes medication (dulaglutide) prior to surgery.

DETAILED DESCRIPTION:
Stress hyperglycemia (SH), defined as a blood glucose >140 mg/dl in hospitalized patients without a prior history of diabetes mellitus (DM) is associated with increased risk of complications and mortality compared to patients with normoglycemia and with known history of DM. Increased counterregulatory hormones (cortisol, glucagon, epinephrine, growth hormone), free fatty acids, inflammation and oxidative stress are likely involved in the pathogenesis of impaired insulin secretion and action leading to stress hyperglycemia. However, no prospective studies have comprehensively examined preoperative glycemic control profiles and their association with the incidence, clinical predictors and underlying mechanisms of SH in general surgical patients. Accordingly, the researchers propose a prospective study investigating clinical, metabolic and inflammatory/oxidative stress biomarker profiles leading to SH. This study will use continuous glucose monitoring (CGM) technology to fully characterize the onset, duration and severity of SH during the perioperative period.

Given the association between stress hyperglycemia and poor hospital outcomes, this study aims to determine if the prevention of stress hyperglycemia is feasible with the single administration of a weekly glucagon-like peptide-1 receptor agonist (GLP-1 RA), a common medication used to treat patients with established diabetes. In addition, the researchers will explore the role of beta-cell function, insulin resistance, and inflammation on the pathogenesis of stress hyperglycemia.

The goals of this study are to: 1) conduct an extensive analysis of preoperative glycemic control and its relationship to clinical, metabolic and biomarker profiles of SH in a high-risk population, and 2) conduct a pilot randomized controlled trial to prospectively determine if single dose use of dulaglutide can improve perioperative glycemic control compared to insulin administration (standard-of-care). Patients qualifying for the study will be approached at their preoperative clinic visit and invited to participate in the prospective observational study arm (Aim 1), and in the interventional trial for prevention of SH with dulaglutide (Aim 2) if they meet inclusion criteria based on oral glucose tolerance testing (OGTT) or lab testing performed for Aim 1. Within 72 hours prior to planned surgery, consented patients will present to the clinical research center (CRC) to undergo evaluation with OGTT and lab testing with CGM placement. Those patients with OGTT or lab results consistent with a diagnosis of prediabetes or newly diagnosed diabetes will be asked if they would like to participate in Aim 2. Patients consenting to participate in Aim 2 will be randomized to receive a subcutaneous injection of dulaglutide 0.75 mg or placebo during the CRC visit, and glycemic control parameters will be followed postoperatively during surgical admission (up to 14 days). In addition to the above, baseline and postoperative levels of serum inflammatory and oxidative stress markers will be obtained to provide further information regarding beta-cell function and insulin resistance in relation to the development of stress hyperglycemia.

ELIGIBILITY:
Inclusion criteria:

* Men and women without known history of diabetes with ages between 45 and 80 years undergoing non-cardiac general or vascular surgery
* BMI ≥30 kg/m2 and pre-DM or DM by OGTT or HbA1c

Exclusion criteria:

* Patients prescribed or taking antihyperglycemic medications
* Patients undergoing cardiac surgery or patients anticipated to require ICU care
* Patients expected to be admitted less than 48-72 hours after surgery
* Severely impaired renal function (eGFR < 30 mL/min) or clinically significant hepatic failure
* Treatment with oral (equivalent to prednisone > 5 mg/day) or injectable corticosteroids
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study; unable to consent
* Pregnant or breast feeding at time of enrollment
* Prisoners
* Patients undergoing gastrointestinal surgery or at high risk for gastrointestinal obstruction/ileus or expected to require gastrointestinal suction
* Patients with delayed gastric emptying, pancreatic or gallbladder disease
* Patients with personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome type 2 (MEN2)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Davis, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Grady Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the publication for this study (including text, tables, figures, and appendices) will be available to other researchers, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available for sharing beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be made available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal. Proposals should be directed to gmdavis@emory.edu. To gain access, data requestors will need to sign a data access/use agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dulaglutide | Placebo
Started | 8 | 8
Completed | 7 | 4
Not Completed | 1 | 4
Not completed — Surgery cancellation | 1 | 2
Not completed — Early discharge (<48 hours) - no CGM data collected | 0 | 1
Not completed — Early discharge (<48 hours) - CGM data collected | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dulaglutide | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Target Glucose Range (70-140 mg/dL) by CGM
Description: The percentage of time in the target glucose range of 70-140 mg/dL, as measured by a continuous glucose monitor (CGM) data was determined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Population: This analysis includes participants with CGM data. One participant who completed the study in the dulaglutide group did not have CGM data available. One participant in the placebo group, who did not complete the study due to being discharged with less than a 48 hour stay, did have CGM data collected and those data are included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 6 | 5
percentage of time | 84.19 (19.70) | 71.82 (27.26)

2. Secondary Outcome: Percentage of Time in Hyperglycemia (Glucose>140 mg/dL)
Description: The percentage of time in hyperglycemia with glucose>140 mg/dL will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

3. Secondary Outcome: Percentage of Time in Hyperglycemia (Glucose>180 mg/dL)
Description: The percentage of time in hyperglycemia with glucose>180 mg/dL will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: Percentage of Time in Hypoglycemia (Glucose <70 mg/dL)
Description: The percentage of time in hypoglycemia with glucose <70 mg/dL will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

5. Secondary Outcome: Percentage of Time in Hypoglycemia (Glucose <54 mg/dL)
Description: The percentage of time in hypoglycemia with glucose <54 mg/dL will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

6. Secondary Outcome: Percentage of Time in Hypoglycemia (Glucose <40 mg/dL)
Description: The percentage of time in hypoglycemia with glucose <40 mg/dL will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

7. Secondary Outcome: Mean Onset of Stress Hyperglycemia During the Postoperative Period
Description: The mean onset time of stress hyperglycemia during the postoperative period by CGM data will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

8. Secondary Outcome: Mean Duration of Stress Hyperglycemia During the Postoperative Period
Description: The mean duration of stress hyperglycemia during the postoperative period by CGM data will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

9. Secondary Outcome: Mean Daily Glucose Values
Description: The mean daily glucose values, as measured by both point of care (POC) glucose testing and CGM data, will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

10. Secondary Outcome: Maximum Daily Glucose Values
Description: The maximum daily glucose values, as measured by both POC glucose testing and CGM data, will be examined.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

11. Secondary Outcome: Perioperative Insulin Requirements
Description: Perioperative insulin requirements will be assessed as the total daily insulin dose.
Time Frame: During hospitalization (up to 5 days postoperatively)
Reporting Status: Not Posted, anticipated posting 2026-05

12. Secondary Outcome: Change in Plasma Cortisol Level
Description: Samples will be collected prior to surgery and 48 to 72 hours after surgery to assess inflammatory and oxidative stress biomarkers.
Time Frame: Baseline, 48 to 72 hours postoperatively
Reporting Status: Not Posted, anticipated posting 2026-05

13. Secondary Outcome: Change in Level of Free Fatty Acids (FFA)
Description: as for outcome 12
Time Frame: Baseline, 48 to 72 hours postoperatively
Reporting Status: Not Posted, anticipated posting 2026-05

14. Secondary Outcome: Change in High Sensitivity C-reactive Protein (hsCRP) Level
Description: as for outcome 12
Time Frame: Baseline, 48 to 72 hours postoperatively
Reporting Status: Not Posted, anticipated posting 2026-05

15. Secondary Outcome: Change in Tumor Necrosis Factor-alpha (TNF-α) Level
Description: as for outcome 12
Time Frame: Baseline, 48 to 72 hours postoperatively
Reporting Status: Not Posted, anticipated posting 2026-05

16. Secondary Outcome: Change in Adiponectin Level
Description: as for outcome 12
Time Frame: Baseline, 48 to 72 hours postoperatively
Reporting Status: Not Posted, anticipated posting 2026-05

17. Secondary Outcome: Change in Level of Thiobarbituric Acid Reactive Substances (TBARS)
Description: as for outcome 12
Time Frame: Baseline, 48 to 72 hours postoperatively
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time that individuals gave consent to participate in the study through the final assessment at hospital discharge, up to 5 days postoperatively.
Arm/Group | Dulaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dulaglutide (N=8) | Placebo (N=8)
Prolonged hospital length of stay due to tachycardia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dulaglutide (N=8) | Placebo (N=8)
Nausea, vomiting, constipation (Gastrointestinal disorders) | 1 | 0
Hypoglycemia, prior to study medication administration (Endocrine disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This clinical trial was performed concurrently with an observational study which will continue until May 2025. Laboratory analysis of samples will be performed after completion of data collection for the observational study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04862234/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT04862234/ICF_001.pdf